CLINICAL TRIAL: NCT02593604
Title: Quality of Life After Wide Surgical Excision in Patients With Hidradenitis Suppurativa
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Fachklinik Hornheide an der Universität Münster (Other)
Responsible Party: Principal Investigator, Tobias Kisch, MD, University Hospital Schleswig-Holstein
Other Study IDs: 14-015; U1111-1176-0162 (Other: WHO)
Record Dates: First submitted 2015-04-11; First posted 2015-11-02 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Hidradenitis Suppurativa; Wide Excision
Keywords: Hidradenitis suppurativa; Wide excision; Quality of Life; Sexual Function
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients undergoing wide surgical excision of their hidradenitis suppurativa areas are asked by telephone about their quality of life by standard questionnaires (WHOQOL-BREF, DLQI, Skindex, MHF, FLQA-d) and their sexual function (FSFI, IIEF).

ELIGIBILITY:
Inclusion Criteria:

* Hidradenitis suppurativa that was wide excised in 2013 in Fachklinik Hornheide
* Agreed to retrospective analysis and questionnaires

Exclusion Criteria:

* Non-compliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hidradenitis suppurativa that were treated in 2013 in Fachklinik Hornheide, Germany, by wide excision of their infected skin areas.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-03-15 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Quality of Life (WHOQOL-BREF) | 2 years postop
  Quality of Life is checked by WHOQOL-BREF
Quality of Life (DLQI) | 2 years postop
  Quality of Life is checked by DLQI
Quality of Life (FLQA-d) | 2 years postop
  Quality of Life is checked by FLQA-d
Quality of Life (Skindex) | 2 years postop
  Quality of Life is checked by Skindex

SECONDARY OUTCOMES:
Sexual Function | 2 years postop
  Sexual Function is checked by IIEF (male) and FSFI (female)
Demographic Parameters | 2 years postop
  Patients' history
Smoking | 2 years postop
  Smoking
Weight and height | 2 years postop
  Weight and height
Wound assessment | 2 years postop
  Localization, Hurley Stage, pain before operation

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kisch, MD, Study Director — University of Schleswig-Holstein, Campus Lübeck, Germany
Locations (1):
- University of Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany